CLINICAL TRIAL: NCT00613860
Title: Sequential Endoscopic Lung Volume Reduction in Patients With Heterogeneous Lung Emphysema
Brief Title: Sequential Endoscopic Lung Volume Reduction
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: complicated patient enrollment
Sponsor: Heidelberg University (Other)
Collaborators: Humboldt-Universität zu Berlin (Other)
Responsible Party: Principal Investigator, Felix JF Herth, CEO, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02/08
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Emphysema; COPD
Keywords: Endoscopic lung volume reduction, heterogeneous emphysema, interventional bronchoscopy
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Zephyr endobronchial valve — Endobronchial valve system to redirect the airflow within the bronchial system

SUMMARY:
Patients with heterogenous emphysema benefits from endoscopic lung volume reduction. Until now the technique is limited to one lobe. In case of collateral ventilation patients show no improvement. Between upper and middle lobe exists the highest collateral flow. The trial examine the hypothesis, that sequential ELVR help especially those patients, which have no benefit after lobar exclusion.

DETAILED DESCRIPTION:
Patients with heterogenous emphysema undergo ELVR, target lobe is the upper lobe right. After 6 weeks the middle lobe will be block too.

Follow-up period 6 months Primary end points: FEV 1, 6-Minute walk test Secondary endpoints. Safety, Symptom scores Number of patients planned 30

ELIGIBILITY:
Inclusion Criteria:

* Heterogenous emphysema
* FEV1 < 45%
* RV > 150%
* TLC > 100%
* TLCO < 40%

Exclusion Criteria:

* Homogeneous emphysema
* Pregnancy
* PCO2 > 50 mmHg

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
FEV 1 6 Minute walk test | 6 months after intervention

SECONDARY OUTCOMES:
Safety Symptom scores | 6 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Felix JF Herth, MD, PhD, Principal Investigator — Thoraxklinik University of Heidelberg
Locations (3):
- Germany (3):
  - Charite, University of Berlin, Berlin
  - Thoraxklinik, University of Heidelberg, Heidelberg
  - Medical Center Nürnberg, Nuremberg

REFERENCES:
- [Background] Strange C, Herth FJ, Kovitz KL, McLennan G, Ernst A, Goldin J, Noppen M, Criner GJ, Sciurba FC; VENT Study Group. Design of the Endobronchial Valve for Emphysema Palliation Trial (VENT): a non-surgical method of lung volume reduction. BMC Pulm Med. 2007 Jul 3;7:10. doi: 10.1186/1471-2466-7-10. PMID 17711594
- [Background] de Oliveira HG, Macedo-Neto AV, John AB, Jungblut S, Prolla JC, Menna-Barreto SS, Fortis EA. Transbronchoscopic pulmonary emphysema treatment: 1-month to 24-month endoscopic follow-up. Chest. 2006 Jul;130(1):190-9. doi: 10.1378/chest.130.1.190. PMID 16840401
- [Background] Venuta F, de Giacomo T, Rendina EA, Ciccone AM, Diso D, Perrone A, Parola D, Anile M, Coloni GF. Bronchoscopic lung-volume reduction with one-way valves in patients with heterogenous emphysema. Ann Thorac Surg. 2005 Feb;79(2):411-6; discussion 416-7. doi: 10.1016/j.athoracsur.2004.07.048. PMID 15680805
- [Background] Yim AP, Hwong TM, Lee TW, Li WW, Lam S, Yeung TK, Hui DS, Ko FW, Sihoe AD, Thung KH, Arifi AA. Early results of endoscopic lung volume reduction for emphysema. J Thorac Cardiovasc Surg. 2004 Jun;127(6):1564-73. doi: 10.1016/j.jtcvs.2003.10.005. PMID 15173708
- [Result] Shah PL, Gompelmann D, Valipour A, McNulty WH, Eberhardt R, Grah C, Egan J, Ficker JH, Wagner M, Witt C, Liebers U, Hopkins P, Gesierich W, Phillips M, Stanzel F, Petermann C, Strange C, Snell G, Herth FJF. Thermal vapour ablation to reduce segmental volume in patients with severe emphysema: STEP-UP 12 month results. Lancet Respir Med. 2016 Sep;4(9):e44-e45. doi: 10.1016/S2213-2600(16)30199-0. Epub 2016 Jul 20. No abstract available. PMID 27451345